CLINICAL TRIAL: NCT00989703
Title: Double Blind, Placebo Controlled, Dose Ranging and Methotrexate Interaction Study for the Assessment of Safety, Tolerability and Pharmacokinetics (PK) of Multiple Oral Doses of GLPG0259 in Healthy Subjects
Brief Title: GLPG0259 Multiple Ascending Dose and Methotrexate Drug-drug Interaction (DDI) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLPG0259-CL-102
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): GLPG0259 25/50/75 mg/day for 14 days
  Interventions: Drug: GLPG0259; Drug: Methotrexate
- 2 (Placebo Comparator): placebo for 14 days
  Interventions: Drug: placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: placebo — oral solution, daily for 14 days
  Arms: 2
Drug: GLPG0259 — oral solution
  Arms: 1
Drug: Methotrexate — 7.5 mg (3 tablets, 2.5 mg/tablet) on study days D-1 and D14
  Other Names: Ledertrexate®

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple increasing oral doses of GLPG0259 compared to placebo.

Also, pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0259 after multiple increasing oral doses, and potential drug-drug interaction with single dose methotrexate will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m², inclusive.

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of oral multiple ascending doses | up to 10 days postdose

SECONDARY OUTCOMES:
Pharmacokinetics of multiple oral doses | up to 10 days postdose
To explore the pharmacokinetic interaction between GLPG0259 and methotrexate (MTX). | up to 10 days postdose
To explore biomarkers of GLPG0259 activity after multiple oral administrations. | up to 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Johan Beetens, PharmD, PhD, Study Director — Galapagos NV; Lien Gheyle, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium